CLINICAL TRIAL: NCT04112303
Title: A Phase 3 Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed-Dose Combination for 12 Weeks in Subjects With Chronic HCV Infection and Compensated Cirrhosis
Brief Title: Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed-Dose Combination for 12 Weeks in Adults With Chronic HCV Infection and Compensated Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-5531; JapicCTI-194989 (Registry Identifier: Japan Pharmaceutical Information Center)
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SOF/VEL (Experimental): Participants received SOF/VEL (400/100 mg) orally once daily for up to 12 weeks.
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — Tablets administered orally once daily
  Other Names: GS-7977/5816; Epclusa®

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of therapy with sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) in adults with chronic hepatitis C virus (HCV) infection and compensated cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic HCV-infected males and non-pregnant/non-lactating females
* Treatment-naïve or treatment-experienced individuals
* Compensated cirrhosis at Screening

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (22):
- Japan (22):
  - Chiba University Hospital, Chiba
  - Fukui-ken Saiseikai Hospital, Fukui
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Hiroshima University Hospital Institution Review Board, Hiroshima
  - Iizuka Hospital, Iizuka
  - Nippon Medical School Hospital, Inzai-shi
  - Saitama Medical University Hospital, Iruma
  - Juntendo University Shizuoka Hospital, Izunokuni
  - Nara Medical University Hospital, Kashihara-shi
  - Toranomon Hospital Kajigaya, Kawasaki-shi
  - Kumamoto Shinto General Hospital, Kumamoto
  - Kurme University Hospital, Kurume-shi
  - Matsuyama Red Cross Hospital, Matsuyama
  - Japanese Red Cross Musashino Hospital, Musashino
  - Hyogo College of Medicine Hospital Institutional Review Board, Nishinomiya
  - National Hospital Organization Nagasaki Medical Center, Omura-shi
  - Osaka Red Cross Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - Osaka University Hospital, Suita-shi
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Toranomon Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Derived] Takehara T, Izumi N, Mochida S, Genda T, Fujiyama S, Notsumata K, Tamori A, Suzuki F, Suri V, Mercier RC, Matsuda T, Matsuda K, Kato N, Chayama K, Kumada H. Sofosbuvir-velpatasvir in adults with hepatitis C virus infection and compensated cirrhosis in Japan. Hepatol Res. 2022 Oct;52(10):833-840. doi: 10.1111/hepr.13810. Epub 2022 Aug 8. PMID 35802063

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Japan. The first participant was screened on 16 October 2019. The last study visit occurred on 25 June 2021.
Pre-assignment Details: 41 participants were screened.
Groups:
- SOF/VEL: Participants received sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) (400/100 mg) tablet orally once daily for up to 12 weeks.
Period: Overall Study
Arm/Group | SOF/VEL
Started | 37
Completed | 36
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of the study drug.
Groups:
- SOF/VEL: Participants received SOF/VEL FDC (400/100 mg) tablet orally once daily for up to 12 weeks.
Arm/Group | SOF/VEL
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 37
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) < Lower Limit of Quantification (LLOQ) 12 Weeks After Discontinuation of Treatment (SVR12)
Description: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) < LLOQ (i.e., 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included all enrolled participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 37
percentage of participants | 100.0 [90.5 to 100.0]
Statistical Analysis 1: Comparison: SOF/VEL; The SVR12 rate was compared to the pre-specified efficacy threshold of 78% using a 2-sided exact 1-sample binomial test at the 0.05 significance level; Test type: Superiority; p < 0.001, 2-sided exact 1-sample binomial test

2. Primary Outcome: Percentage of Participants Who Experienced Any Treatment-Emergent Adverse Event (TEAE) Leading to Discontinuation of Study Drug
Description: TEAEs were defined as any AEs with an onset date on or after the study drug start and no later than 30 days after permanent discontinuation of study drug and/or any AEs leading to premature discontinuation of the study drug.
Time Frame: First dose date up to Week 12.1
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 37
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at 4 Weeks After Discontinuation of Treatment (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ (i.e.15 IU/mL) at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 37
percentage of participants | 100.0 [90.5 to 100.0]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at 24 Weeks After Discontinuation of Treatment (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ (i.e.15 IU/mL) at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 37
percentage of participants | 100.0 [90.5 to 100.0]

5. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IL/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment.
Time Frame: First dose date up to posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 37
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment to Posttreatment Week 24; Adverse Events: First dose date up to Week 12.1 plus 30 days
Description: All-Cause Mortality: All Enrolled Analysis Set included all participants who received a study subject identification number in the study after screening. Adverse Events: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | SOF/VEL
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 5/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=37)
Patella fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=37)
Diarrhoea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT04112303/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT04112303/SAP_001.pdf